CLINICAL TRIAL: NCT04753229
Title: Comparison of the Ki67 Proliferation Index of Pancreatic Neuroendocrine Neoplasia Between Preoperative Micro-biopsies and Surgical Specimens
Brief Title: Ki67 Proliferation Index of Pancreatic Neuroendocrine Neoplasia
Acronym: TNE-P-Ki
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: TNE P Ki-IPC 2020-046
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Neuroendocrine Tumors
Keywords: pancreatic neuroendocrine tumor; Ki67; artificial intelligency
MeSH Terms: conditions — Neuroendocrine Tumors; Adenoma, Islet Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective, monocentric study involving 50 patients with pancreatic neuroendocrine neoplasia resected between January 2008 and June 2020 at Paoli Calmettes Institute.

The primary objective of the study is to evaluate the grade concordance rate, based on Ki67 obtained on the pre-operative micro-biopsy and the surgical specimen.

Based on the histology slides obtained in the course of the treatment, several Ki67 recounts will be performed on pre-operative tumor micro-biopsies and on tumors resected after surgery:

* a manual count (on photo printed in the hotspot area according to World Health Organization (WHO) 2017 recommendations, by an expert pathologist and a junior pathologist.
* Automated counting using specific software based on artificial intelligence (Qpath software).

On the other hand, clinical, surgical and anatomopathological data will be collected in order to follow the patient evolution.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resection of pancreatic neuroendocrine neoplasia by surgery at Paoli Calmettes Institute between January 2008 and June 2020
* Patients who had a pre-surgical evaluation of Ki67 on micro-biopsy equipment obtained by echo-endoscopy.

Exclusion Criteria:

* Patient with a mixed tumor of the pancreas.
* Patient with a pancreas tumor composed of several nodules of similar size without a main mass and for which it is not possible to determine the biopsied nodule during echo-endoscopy.
* Initial micro-biopsy in a private pathology laboratory
* Initial subechoendoscopic puncture cytology only (Ki67 not possible)
* No initial micro-biopsy and surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had a pre-surgical evaluation of Ki67 on micro-biopsy equipment obtained by echo-endoscopy and a resection of pancreatic neuroendocrine neoplasia by surgery at Paoli Calmettes institute between January 2008 and June 2020
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Ki67 Grade | on pre-operative micro-biopsies
  Evaluation by a pathologist by manual counting according to WHO 2017 recommendations
Ki67 Grade | on surgical specimens
  Evaluation by a pathologist by manual counting according to WHO 2017 recommendations

SECONDARY OUTCOMES:
Percentage of Ki67 positive cells on total counted cells | on preoperative micro-biopsies
  Evaluation by a pathologist by manual counting according to WHO 2017 recommendations
Percentage of Ki67 positive cells on total counted cells | on surgical specimens
  Evaluation by a pathologist by manual counting according to WHO 2017 recommendations
Percentage of Ki67 positive cells on total counted cells | on preoperative micro-biopsies
  Evaluation by digital pathology before and after machine learning
Percentage of Ki67 positive cells on total counted cells | on surgical specimens
  Evaluation by digital pathology before and after machine learning

CONTACTS AND LOCATIONS:
Overall Officials: Flora Poizat, Principal Investigator — Institut Paoli-Calmettes (IPC)